CLINICAL TRIAL: NCT01913860
Title: Supporting the Improvement and Management of Prescribing for Urinary Tract Infections (SIMPle): Protocol for a Randomised Complex Intervention
Brief Title: Supporting the Improvement and Management of Prescribing for Urinary Tract Infections (SIMPle)
Acronym: SIMPle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Akke Vellinga, Senior Lecturer Primary Care, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ICE/2011/10
Record Dates: First submitted 2013-07-26; First posted 2013-08-01 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Uncomplicated Urinary Tract Infection
Keywords: UTI; antibiotics; prescribing; primary care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Control group will receive usual care
- Improve GP prescribing behaviour (Active Comparator): Improve GP prescribing behaviour will be promoted through personalised audit and feedback reports, delivered through face to face workshops within practice.
  Interventions: Behavioral: Improving GP antibiotics prescribing behaviour
- Improved delayed GP prescribing (Active Comparator): Improved delayed GP prescribing will be promoted through the antibiotic prescribing guidelines and personalised audit and feedback reports. Additional scientific evidence will be provided related to delayed prescribing.
  Interventions: Behavioral: Improving GP antibiotics prescribing behaviour

INTERVENTIONS:
Behavioral: Improving GP antibiotics prescribing behaviour — GPs will be asked to code their UTI patients within their patient management software. Anonomysed coded patients will be electronically extracted and this information will be provided as an audit and feedback report of the GPs antibiotic prescribing practices.
  Arms: Improve GP prescribing behaviour; Improved delayed GP prescribing

SUMMARY:
Background The over use of antimicrobials is recognised as the main selective pressure driving the emergence and spread of antimicrobial resistance in human bacterial pathogens. Urinary Tract Infections (UTIs) are one of the most common infections presented in primary care and empirical antimicrobial treatment is currently recommended. Previous research has identified that a substantial proportion of Irish GPs prescribe antimicrobials for UTI that are not in accordance with the Guidelines for Antimicrobial Prescribing in Primary Care in Ireland.

Aim To design, implement and evaluate the effectiveness of a complex intervention on GP antimicrobial prescribing and adult (18 years of age and over) patients' antimicrobial consumption when presenting with a suspected UTI.

Methods The SIMPLE study is a randomised three armed intervention with practice level randomisation. Adult patients presenting with suspected UTI in primary care will be included in the study.

The intervention integrates components for both GPs and patients. For GPs the intervention includes interactive workshops, audit and feedback reports and automated electronic prompts summarising recommended first line antimicrobial treatment and, for one intervention arm, a recommendation to consider delayed antimicrobial prescribing. For patients multimedia applications and information leaflets are included. A minimum of 920 patients will be recruited through 30 practices. The primary outcome is change in prescribing of first line antimicrobials in accordance with the Guidelines for Antimicrobial Prescribing in Primary Care in Ireland. The intervention will take place over 15 months. Data will be collected through a remote electronic anonymised data extraction system (iPCRN), a text messaging system and through GP and patient interviews and surveys. The intervention will be strengthened by the implementation of a social marketing framework and an economic evaluation.

DETAILED DESCRIPTION:
Today, 80% of antimicrobial prescribing takes place in the community by general practitioners (GPs). Ireland is one of only three countries in Europe where the level of outpatient antimicrobial prescribing is increasing. Within this context, the inappropriate and overprescription of antimicrobials by GPs is a recognized factor contributing to the spread of AMR. The Guidelines for Antimicrobial Prescribing in Primary Care in Ireland provide advice on the selection of antimicrobial drugs for common infections and recommend the use of specific antimicrobials, with reserved drugs for more serious infections. However, despite the widespread availability of these guidelines, recent research has identified that less than 40% of outpatient prescriptions for urinary tract infections (UTIs) are made out according to first-line recommendations.

Urinary tract infections are predominantly caused by a bacteria; Escherichia coli, and are generally treated empirically, prior to the results of antimicrobial susceptibility testing. Antimicrobial resistance is now a critical factor in the treatment of UTIs, the second most common bacterial infection in primary care.

Social marketing is the conceptual framework that guided the development of this intervention. Formative (qualitative) research explored the culture of antimicrobial prescribing from both the GP's and the patient's perspective. Through a series of interviews with GPs (n = 15) and focus groups with patients (n = 35), the predictors of a GP's decision to prescribe an antimicrobial and the patient's expectation to receive an antimicrobial were explored.

The aim of SIMPle was to design, implement and evaluate the effectiveness of a complex intervention on GP antimicrobial prescribing and adult (18 years of age and over) patients' antimicrobial consumption when presenting with a suspected UTI. The primary outcome was to increase the number of first-line antimicrobial prescriptions, as recommended in the Guidelines for Antimicrobial Prescribing in Primary Care in Ireland (2011), for suspected UTIs in primary care by 10% in adult patients.

Methods The cluster for this intervention is the practice, and all GPs within each practice will be invited to participate. The baseline population for recruitment of patients will be formed by all practices in the West of Ireland who submit urine samples to the Galway University Hospitals (GUH) laboratory. The most popular patient management software system was chosen, because the SIMPle study builds on remote data extraction, the provision of audit and feedback reports and computer prompts integrated within the GP's patient management software system. This study will be undertaken in four phases: Phase 1, baseline data collection; Phase 2, GP intervention; Phase 3, patient intervention and Phase 4, endpoint data collection. Computerized remote data extraction is facilitated by the Irish Primary Care Research Network (iPCRN) and patient data are identified through the appropriate coding of suspected UTI consultations in the patient management software system. To promote and encourage consultation coding, which is currently not routine practice, the intervention will be preceded by a coding workshop at the beginning of Phase 1. All practices will be required to register with the iPCRN during or before the coding workshop. Practices will be monitored for two months after the delivery of the workshop to establish uptake of coding, whilst also facilitating a baseline data collection period (Phase 1). Phase 2 will begin with an interactive workshop (intervention arms A and B), which will introduce the intervention components specific to each arm. Phase 3 will see the roll-out of the patient education in all of the practices. The antimicrobial prescribing within each practice will be monitored for six months during Phases 2 and 3 through audit and feedback reports. Evaluation of the impact of the intervention will be carried out in Phase 4.

All patients are eligible if aged 18 years and over and presenting with symptoms of an UTI, as determined by the GP through the consultation coding.

Previous research has established that 56% of UTI patients receive an antimicrobial, with only 38% of prescription made out for the recommended first-line treatment.

Sample size calculations are based on an absolute 10% increase in first-line prescriptions according to guidelines (primary outcome). Additional assumptions for sample size calculations include power of 80% and α of 5%, Practice attrition is dependent on the completeness of consultation coding, which will be monitored and corrected during Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients presenting with a suspected urinary tract infection to their general practitioner (GP)

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2577 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Relative number of prescriptions of first line antimicrobials | 3 and 9 months
  Increase in the relative number of prescribing (over all UTI consultations) of first line antimicrobials as recommended in the Guidelines for Antimicrobial Prescribing in Primary Care in Ireland (2010), for suspected UTI in primary care by 10% in adult patients.

SECONDARY OUTCOMES:
Relative number of antimicrobial prescriptions for UTI | 3 and 9 months
  To compare the effect of the intervention on the frequency of antimicrobial prescribing and antimicrobial consumption in patients presenting with an UTI
Number of delayed prescriptions for UTI | 3 and 9 months
  To measure the uptake delayed antimicrobial prescribing for UTI and the impact of this treatment approach on UTI GP reconsultation visits.

OTHER OUTCOMES:
relative change in beliefs | 0 and 9 months
  To assess a change in cognitive beliefs (knowledge and attitudes) of GPs related to antimicrobial prescribing with qualitative survey
Cost of intervention | 9 months
  conduct a cost-effectiveness evaluation of the SIMPle intervention
Relative change in prescribing rates | 9 months
  compare the prescribing rates of the intervention arms with regional UTI antimicrobial prescribing rates

CONTACTS AND LOCATIONS:
Overall Officials: Akke Vellinga, PhD, Study Director — NUI Galway; Andrew W Murphy, MD, Principal Investigator — NUI Galway
Locations (1):
- NUI Galway, Galway, Galway, Ireland

REFERENCES:
- [Derived] Duane S, Tandan M, Murphy AW, Vellinga A. Using Mobile Phones to Collect Patient Data: Lessons Learned From the SIMPle Study. JMIR Res Protoc. 2017 Apr 25;6(4):e61. doi: 10.2196/resprot.6389. PMID 28442451
- [Derived] Duane S, Domegan C, Callan A, Galvin S, Cormican M, Bennett K, Murphy AW, Vellinga A. Using qualitative insights to change practice: exploring the culture of antibiotic prescribing and consumption for urinary tract infections. BMJ Open. 2016 Jan 11;6(1):e008894. doi: 10.1136/bmjopen-2015-008894. PMID 26754175
- [Derived] Tandan M, Duane S, Vellinga A. Do general practitioners prescribe more antimicrobials when the weekend comes? Springerplus. 2015 Nov 24;4:725. doi: 10.1186/s40064-015-1505-6. eCollection 2015. PMID 26636013
- [Derived] Vellinga A, Galvin S, Duane S, Callan A, Bennett K, Cormican M, Domegan C, Murphy AW. Intervention to improve the quality of antimicrobial prescribing for urinary tract infection: a cluster randomized trial. CMAJ. 2016 Feb 2;188(2):108-115. doi: 10.1503/cmaj.150601. Epub 2015 Nov 16. PMID 26573754
- [Derived] Duane S, Callan A, Galvin S, Murphy AW, Domegan C, O'Shea E, Cormican M, Bennett K, O'Donnell M, Vellinga A. Supporting the improvement and management of prescribing for urinary tract infections (SIMPle): protocol for a cluster randomized trial. Trials. 2013 Dec 23;14:441. doi: 10.1186/1745-6215-14-441. PMID 24359543
- See also: Simple Study website — http://simple.nuigalway.ie/